CLINICAL TRIAL: NCT03736187
Title: Combination Vs Single Antibiotics for Prevention of SSI in Obese Women Undergoing CS
Brief Title: Antibiotics for Prevention of SSI in Obese Women Undergoing CS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abeer mohammed abd allah elsayed, Cairo governorate,hadaik elqoba,elkhalig elmasry street, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Antibiotics for SSI
Record Dates: First submitted 2018-03-27; First posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cephalexin; Metronidazole

STUDY DESIGN:
Intervention Model Description: 2 Groups of obese women under elective cesarean section
Who Masked: Participant
Masking Description: Two equal groups,140 women in each group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cephalexin (Experimental): Group a will receive cephalexin 1gm before skin incision intravenous
  Interventions: Drug: Cephalexin
- Cephalexin &metronidazole (Experimental): Group b will receive cephalexin 1gm intravenous plus 1gm metronidazole rectally before skin incision
  Interventions: Drug: Cephalexin

INTERVENTIONS:
Drug: Cephalexin — Giving cephalexin and metronidazole in one group &cephalexin alone in another group
  Other Names: Metronidazole

SUMMARY:
Effect of cephalexin plus metronidazole on SSI better than cephalexin alone in obese women undergoing CS

DETAILED DESCRIPTION:
Comparison between efficacy of cephalexin alone and cephalexin plus metronidazole on surgical site infection in obese women undergoing CS and follow up of any signs of wound infection

ELIGIBILITY:
Inclusion Criteria:

* obese women under elective CS

Exclusion Criteria:

* immunodeficient women

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Wound infection | One week
  Fever, redness, ecchymosis and tenderness

IPD SHARING:
Plan to Share IPD: Undecided